CLINICAL TRIAL: NCT06720376
Title: Assessment of Spondyloarthritis in an Acute Anterior Uveitis Inception Cohort: a Cross Sectional and Prospective Comparative Study of HLA-B27-positive and -negative Cases
Brief Title: Observational Prospective Turkish Inception Cohort of Uveitis and Spondyloarthritis
Acronym: OPTICUS
Status: Recruiting | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Mehmet Pamir Atagunduz, Professor, Marmara University
Other Study IDs: OPTICUS.001
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Spondylarthritis; Uveitis, Anterior
Keywords: Spondylarthritis, Acute Anterior Uveitis, Inflammatory Back Pain, HLA-B27
MeSH Terms: conditions — Spondylarthritis; Uveitis, Anterior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — As the first stage, blood samples will be collected in EDTA tubes, subsequently will be isolated with commercial kits. DNA samples will be stored at -80 fridge.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- main cohort

SUMMARY:
Spondyloarthritis (SpA) encompasses a group of inflammatory rheumatic diseases characterized by axial and/or peripheral arthritis, along with extra-articular manifestations such as enthesitis, dactylitis, uveitis, and skin lesions. Axial spondyloarthritis (axSpA), the hallmark of which is chronic sacroiliitis, can progress to vertebral fusion ("bamboo spine") in advanced cases. The prevalence of axSpA varies globally, ranging from 0.1% to 1.4%, with a higher incidence in men and a typical onset in the second or third decades of life. Diagnostic approaches include imaging techniques such as sacroiliac MRI and radiographs, alongside clinical criteria like inflammatory back pain, NSAID responsiveness, peripheral arthritis, and HLA-B27 positivity. Disease management primarily involves NSAIDs, with biologics used for refractory cases, and disease activity is monitored using indices such as BASDAI and ASDAS.

Acute anterior uveitis (AAU) is the most common extra-articular manifestation of SpA, particularly associated with HLA-B27 positivity. It often presents unilaterally with redness, pain, and photophobia but can lead to severe complications if inadequately treated. Around 50% of patients with HLA-B27-positive AAU have underlying SpA, and the prevalence of uveitis increases with longer disease duration. While the link between SpA and AAU is well-established, further research is needed to determine optimal systemic treatment and follow-up protocols. This study aims to assess the prevalence and clinical characteristics of SpA in patients presenting with AAU at ophthalmology clinics.

ELIGIBILITY:
Inclusion Criteria:

* patients with uveitis

Exclusion Criteria:

* patients diagnosed spondyloarthiritis before from the uveitis attack
* patients with infectious uveitis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Turkish population
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-01-15 (Actual); Primary Completion 2028-01-15 (Estimated); Study Completion 2030-01-15 (Estimated)

PRIMARY OUTCOMES:
Assesing the Prevalance of Axial- and Peripheral Spondyloarthritis according to ASAS Classification Criteria among Patients with Acute Anterior Uveitis. | Cross-sectional anaylsis of the first two hundered patients for the prevalance of Spondyloarthritis is anticipated to be analyzed at the end of the second year after the inclusion of the first patient with acute anterior uveits.
  Presence of undiagnosed or known Spondyloarthritis will be assessed in a cross-sectional manner at time of acute anterior uveitis.
Assesing the Incidence of Axial- and Peripheral Spondyloarthritis according to ASAS Classification Criteria among Patients with Acute Anterior Uveitis after first diagnosis. | Cross-sectional anaylsis of the first two hundered patients for the prevalance of Spondyloarthritis is anticipated to be analyzed at the end of the fifth year after the inclusion of the last patient with acute anterior uveits.
  Development of an full-blown Spondyloarthritis will be assessed long-term in a prospective manner.

SECONDARY OUTCOMES:
Comparison of the HLA-B27 status among acute anterior uveitis patients with and without spondyloarthritis. | Cross-sectional anaylsis of the first two hundered patients for the prevalance of HLA-B27 is anticipated to be analyzed at the end of the second year after the inclusion of the first patient with acute anterior uveits.
  HLA-B27 status will be assessed in patints with idiopathic acute- and spondyloarthritis associated anterior uveitis will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University School of Medicine, Istanbul, Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code